CLINICAL TRIAL: NCT00570440
Title: Continuous Versus Cyclic Use of Combined Oral Contraceptive Pills
Brief Title: Continuous Use of COCs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: La Asociación Pro Bienestar de la Familia de Guatemala (APROFAM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9964
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Pregnancy Prevention
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Ethinyl Estradiol; Levonorgestrel

ARMS (2):
- A (Experimental)
  Interventions: Drug: Oral contraceptives--ethinyl estradiol, levonorgestrel
- B (Active Comparator)
  Interventions: Drug: Oral contraceptives--ethinyl estradiol, levonorgestrel

INTERVENTIONS:
Drug: Oral contraceptives--ethinyl estradiol, levonorgestrel — 3 visits - screening/enrollment, 6-months and 12 months

SUMMARY:
The primary objective is to determine if continuous COC use leads to higher continuation rates over 12 months of follow up than use of the standard 28-day COC regimen.

DETAILED DESCRIPTION:
Family Health International has recently initiated a USAID funded study to investigate the pregnancy rates, continuation rates, and acceptability of COCs in women taking COCs by the 21/7 cyclic regimen compared with the continuous use of COCs with bleeding-signaled hormone-free intervals. The primary objective is to determine whether continuous COC use leads to higher 12-month continuation rates than use of the standard 28-day COC regimen. Secondary objectives are to 1) compare pregnancy probabilities through 6 and 12 months between the continuous use group and the 28-day group 2) compare COC continuation rates through 6 months between the continuous use group and the 28-day group 3) compare acceptability of the two COC regimens 4) to compare bleeding and other side effects between the continuous use group and the 28-day group 5) to compare hemoglobin/hematocrit between the continuous use group and the 28-day group

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Currently has menstrual periods every 21-35 days
* Willing and able to be randomly assigned to one of the two study groups and to comply with all study requirements
* Has signed the informed consent form
* Has a negative urine pregnancy test at enrollment

Exclusion Criteria:

* Has contraindications to COC use (see WHO MEC-3rd edition)
* Is in any other research study
* Has been pregnant in the past 3 months
* Is breastfeeding or has breastfed in the past 3 months
* Is currently using an IUD (women who agree to IUD removal are eligible once the IUD is removed)
* Has had an injection of DMPA in the past 6 months
* Has had an injection of NET-EN in the past 3 months
* Has used combined injectables, oral contraceptive pills, implants, or a hormonal IUD in the past 2 months
* Has had any of the following conditions since her last pregnancy, or since menarche if never pregnant:

  * Pelvic infection treated with antibiotics
  * Diagnosis of infertility
  * Endometriosis

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 362 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
12 month cumulative COC discontinuation probabilities | 12 months

SECONDARY OUTCOMES:
Pregnancy rates through 6 and 12 months; 6 month cumulative discontinuation probabilities; acceptability; bleeding and other side effects; hemoglobin/hematocrit | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Nanda, MD, MHS, Principal Investigator — FHI 360
Locations (2):
- PROFAMILIA - Santo Domingo, Dominican Republic, Ens. Luperon, Santo Domingo Province, Dominican Republic
- PROFAMILIA - Managua, Nicaragua, Managua, Managua Department, Nicaragua

REFERENCES:
- [Derived] Nanda K, Lendvay A, Kwok C, Tolley E, Dube K, Brache V. Continuous compared with cyclic use of oral contraceptive pills in the Dominican Republic: a randomized controlled trial. Obstet Gynecol. 2014 May;123(5):1012-1022. doi: 10.1097/AOG.0000000000000235. PMID 24785854